CLINICAL TRIAL: NCT06831110
Title: Using Aquagenic Wrinkling to Predict CF Carrier State
Brief Title: Aquagenic Wrinkling Prediction
Status: Recruiting | Type: Observational
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Philip Polgreen, Professor, University of Iowa
Other Study IDs: 202410028
Record Dates: First submitted 2025-02-05; First posted 2025-02-17 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Aquagenic Wrinkling of Palms; Carrier State

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Potential Cystic Fibrosis Carriers: Participants that are identified as potential cystic fibrosis carriers based on aquagenic wrinkling results.
  Interventions: Procedure: Aquagenic Wrinkling
- Potential Controls: Participants that are identified as potential controls based on aquagenic wrinkling results.
  Interventions: Procedure: Aquagenic Wrinkling

INTERVENTIONS:
Procedure: Aquagenic Wrinkling — Participants will be asked to remove all jewelry from the hand(s) and wrist(s) that will be undergoing the aquagenic wrinkling procedures. Photographs will be taken of the palmar surface of the hand(s). The participant will submerge the hand(s) undergoing testing in a water bath for one minute. After one minute, they will remove their hand(s), dry them gently with a towel, and photographs will be taken of the palmar surface of the hand(s). The participant will re-submerge their hand(s) in the appropriate conditions for another minute and the process will be repeated 20 times for 20 total minutes submerged in the water.

SUMMARY:
The goal of this observational study is to determine whether an aquagenic wrinkling procedure (i.e., soaking hands in a water bath for up to 20 minutes) can be used as a screening tool for cystic fibrosis carrier status.

Participants will complete one visit where they will undergo an aquagenic wrinkling procedure to see how their hands respond.

ELIGIBILITY:
Inclusion Criteria:

* Interested in participating in other CF Carrier-related research studies.

Exclusion Criteria:

* CF patient status
* Unable to speak English
* Unable to provide written informed consent
* Prisoner status
* An open wound on either hand
* A tattoo on either hand
* Missing any portion of either hand
* Diagnosis of Diabetes
* Diagnosis of Hyperhidrosis
* Diagnosis of Raynaud's Disease
* Diagnosis of Atopic Dermatitis
* Regularly taking ACE inhibitors or angiotensin receptor blockers

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: University students
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Human Observation of Wrinkling | Up to 20 minutes
  Photos of hands will be scored on a scale of 0 (no wrinkling) to 4 (severe wrinkling) at each minute by human observers.
Machine-Learning Observation of Wrinkling | Up to 20 minutes
  Photos of hands will be scored by a machine-learning algorithm at each minute.

CONTACTS AND LOCATIONS:
Overall Officials: Philip M Polgreen, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No